CLINICAL TRIAL: NCT05042492
Title: Postoperative Oedema Management Following Neuromuscular Electro- Stimulation of the Peroneal Nerve Using the gekoTM Device After Total Knee Arthroplasty
Brief Title: The Post-operative Effect on Formation of Oedema After Total Knee Arthroplasty With or Without the Use of a Nerve Stimulator (the gekoTM Device)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: moveUP bv (Industry)
Collaborators: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MMS.2020.058
Record Dates: First submitted 2021-01-08; First posted 2021-09-13 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Knee; Edema Leg; Joint Diseases; Rehabilitation
Keywords: Total Knee Arthroplasty; Osteoarthritis; Arthritis; Edema; Patient reported outcomes (PROMs); Telerehabilitation; Physiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Joint Diseases; Osteoarthritis; Arthritis; Edema

STUDY DESIGN:
Intervention Model Description: The study was designed as a single centre, prospective, randomised (1:1), dual arm, single treatment, unblinded, interventional study that will be performed on patients undergoing unilateral TKA for primary OsteoArthritis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: SC (moveUP) (No Intervention): In group 1: moveUP (class 1, CE-marked, medical device) is being used as the rehabilitation solution after TKA. It has become a valid digital rehabilitation solution and is recognised by the Belgian government as mobile health application in rehabilitation of hip and knee arthroplasty surgeries. It's a full service with daily personalized and individualized follow up by certified physical therapists and certified health care providers. The use of tele-rehabilitation for TKA patients has been internationally recognized with the 2018 John N. Insall Award during the American Knee Society Meeting
- Group 2: SC (moveUP) with 10 days of geko (Experimental): In group 2: Next to SC (moveUP), the application of a single gekoTM device is used on the operated leg after surgery (day 0). This device will be worn for 24 hours and at least 8 hours from day 1 until day 10.
  Interventions: Device: gekoTM

INTERVENTIONS:
Device: gekoTM — The gekoTM device is a small, transcutaneous nerve stimulator that is placed non-invasively on the skin, whereby the surface electrodes will be attached close to the peroneal nerve. Activation of the peroneal nerve causes contraction of the calf muscle pump, which will increase blood circulation that corresponds to 60% of walking. The increased blood circulation reduces the pressure difference between capillaries and the surrounding tissue and transfers the tissue fluid back into the veins and lymph fibers
  Arms: Group 2: SC (moveUP) with 10 days of geko

SUMMARY:
This study will investigate whether the recovery of muscle function of total knee arthroplasty is accelerated with the use of the gekoTM device along with its effect on reducing symptoms such as oedema and inhibition of the muscle function.

DETAILED DESCRIPTION:
This study will investigate total knee arthroplasty patients:

* One group gets standard of care (i.e. performing exercises & guidance by a physiotherapist via a CE-marked mobile application, called moveUP)
* Second group gets standard of care + GekoTM device (i.e. non-invasive neuromuscular electrostimulation applied at the peroneal nerve for 10 days after the operation date.)

The primary objective of the study is to assess the post-operative effect of gekoTM on formation of oedema (measured by perometer).

The effect of the gekoTM device on the muscle function & the overall recovery will be also investigated.

To collect parameters, the patient will be asked to complete questionnaires, including the following patient reported outcomes (PROMs): Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Society Score (KSS), Euroqol Health questionnaire EQ5D, Forgotten Joint Score (FJS), Oxford Knee Score (OKS).

The collection of the PROMs will give an indication on outcome and overal recovery in the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Primary TKA planned for degenerative OA
* Subjects must be discharged to home environment and be able to independently perform the activities of daily life
* Obtain a written informed consent

Exclusion Criteria:

* TED stockings, Dauerbinde, other compressive bandages
* Mechanical foot pump
* Cooling device type 'Game Ready'
* Posttraumatic OA of the knee
* History of DVT / Flebitis / Pulmonary embolism
* Surgical treatment of venous insufficiency <1y prior to TKA surgery
* Neurological deficit of lower limbs
* Current sciatic irradiating pain in lower limbs
* History of lumbar fusion
* Knee Arthroscopy of the involved limb <6m prior to TKA surgery
* Any per-operative complication related to the TKA procedure (bleeding, fracture, vascular injury, cardiac complication, pulmonary complication)
* In case of a release during the TKA procedure
* Any per-operative (e.g. epidural catheter, urethral catheter, intra articular catheter) or post-operative procedure that might interfere with the rehabilitation during and after hospitalization
* Any scheduled surgery in the 3 months following the reference surgery;
* Any significant medical condition (e.g. Parkinson's disease, multiple sclerosis, cerebral vascular accident) that might interfere with the rehabilitation
* Any significant psychiatric disorders, active alcohol/drug abuse
* Subject is either pregnant or interested in becoming pregnant during the duration of the study
* Subjects who are currently involved in any investigational drug or device study or have been enrolled in such study within the last 3 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to assess the post-operative effect of gekoTM on formation of oedema following Total Knee Arthroplasty (TKA) | until end of rehabilitation (+- 3 months after TKA operation)
  This is measured by the use of a perometer. For each patient, change in limb volume shall be calculated as a percentage of original limb volume.
  Shapiro-Wilk test shall be used to test whether there is a significant (p<0.05) departure from normal distribution in either group.

SECONDARY OUTCOMES:
Incidence of Adverse Events | until end of rehabilitation (+- 3 months after TKA operation)
  Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs, including an abnormal laboratory finding, in subjects, users or other persons, in the context of a clinical investigation, whether or not related to the investigational device.
  (MDR Article 2(57)). The total number adverse events and the total number (%) of patients that had at least 1 adverse event will be stated.
Incidence of Device Deficiency | during 10 days after TKA operation
  Any inadequacy in the identity, quality, durability, reliability, safety or performance of an investigational device, including malfunction, use errors or inadequacy in information supplied by the manufacturer.(MDR Article 2(59))
Oedema measurements - subjective slider | until end of rehabilitation (+- 3 months after TKA operation)
  Temperature/swelling: Identical subjective slider as daily evaluated by the patient itself presenting the result as a Visual Analog Scale score, minimum 0 (no swelling) maximum 100 (Very swollen)
Oedema measurements - photographic evaluation | until end of rehabilitation (+- 3 months after TKA operation)
  picture of both knees (moveUP): Patients need to make a picture of both knees, using the photo camera on their smartphone to see the swelling of the operated leg compared to the non-operated leg and to evaluate the swelling of the operated leg.
  This blind assessment of pictures is performed by a physical therapist.
Patient Reported Outcome Measures (PROM's) | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
  The PROMS's measured:
  - KOOS: Knee injury and Osteoarthritis Outcome Score for Joint Replacement. 42 items on 5-point Likert scale (multiple choice), total score is on 100, lower scores being indicative of worse knee conditions and higher scores being indicative of better knee condition
Patient Reported Outcome Measures (PROM's) | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
  The PROMS's measured:
  - KSS: Knee Satisfaction Score. Multiple choice scale. Total score on 100, lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.
Patient Reported Outcome Measures (PROM's) | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
  The PROMS's measured:
  - EQ5-D: Euroqol Health questionnaire. 5 items on 5-point Likert scale (multiple choice). Total score on 100. Secondly there is also 1 visual analog scale (VAS). The VAS Score is scored separately with lower scores being indicative of worse health and higher scores being indicative of better health (generic questionnaire, not disease specific)
Patient Reported Outcome Measures (PROM's) | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
  The PROMS's measured:
  - OKS: Oxford Knee Score. 12 items Multiple choice. a lower score can be indicative for bad function or pain after TKA
Patient Reported Outcome Measures (PROM's) | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
  The PROMS's measured:
  - FJS: Forgotten Joint score. 12-item mutiple choice score. Total score on 100 (%), lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.
Pain level | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
  Visual analogue scale (VAS), a 0-100 scale with 100 score = the worst pain the patient can feel and 0 = the patient feels no pain
Number of days of Painkiller intake | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
  PK intake stop is defined as no PK consumption for 3 consecutive days with no new 3 day-period of PK intake.
Dosage Painkiller intake | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
Number of days of NSAID intake | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
  NSAID intake stop is defined as no NSAID consumption for 3 consecutive days with no new 3 day-period of NSAID intake.
Dosage NSAID intake | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
Sleep duration | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
  the wearable measures accelerations during 23h-8h and gives an assumption duration of sleep during the night. The assumption of amount of sleep is based on: very little registration (deep sleep), little movements (light sleep), a lot of movements (waking up).
Sleep quality | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
  the wearable measures accelerations during 23h-8h and gives an assumption quality of sleep during the night. The assumption of amount of sleep is based on: very little registration (deep sleep), little movements (light sleep), a lot of movements (waking up).
Recovery of physical activity (PA) | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
  number of weeks until post-operative PA level is similar to pre-operative PA level, meaning there is no significant difference between mean post-operative step count (calculated on each post-operative week) and mean pre-operative step count (calculated on 7 days before surgery).
Number of days of crutches use | until end of rehabilitation (+- 3 months after TKA operation)
Resume driving a car | until end of rehabilitation (+- 3 months after TKA operation)
  Number of days post-operative
Overall Net Promotor Score (NPS) of the rehabilitation in general | 2 weeks pre-operative until end of rehabilitation (+- 3 months after TKA operation)
  NPS = How likely would you recommend the rehabilitation to your friends or family?". Visual analogue scale (VAS), a 0-100 scale with 100 score = very likely and 0 = not likely
Satisfaction and feedback on the geko device (only for patients using the geko) | during 10 days after TKA operation
  Including:
  * Ease of use
  * Required level of stimulation (1 to 11)
  * Adherence to the geko use: daily collection of number of hours worn during the 10 days the geko device is used

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Van Overschelde, Study Director — Algemeen Ziekenhuis Maria Middelares
Locations (1):
- AZ maria middelares, Ghent, East-Flanders, Belgium